CLINICAL TRIAL: NCT02750761
Title: A Phase 1, Single-Administration Pharmacokinetic and Safety Study of Oral and IV Tedizolid Phosphate in Hospitalized Subjects 2 to <12 Years Old
Brief Title: A Study of Oral and Intravenous (IV) Tedizolid Phosphate in Hospitalized Participants, Ages 2 to <12 Years, With Confirmed or Suspected Bacterial Infection (MK-1986-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1986-013; TR701-120 (Other: Cubist Protocol Number); 2015-004595-29 (EudraCT Number); MK-1986-013 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-04-01; First posted 2016-04-25 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Gram-Positive Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — tedizolid phosphate; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 years) (Experimental): Participants 6 to <12 years of age received a single intravenous infusion of tedizolid phosphate dosed at 5 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
  Interventions: Drug: Tedizolid Phosphate (IV)
- Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 years) (Experimental): Participants 6 to <12 years of age received a single intravenous infusion of tedizolid phosphate dosed at 4 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
  Interventions: Drug: Tedizolid Phosphate (IV)
- Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 years) (Experimental): Participants 2 to <6 years of age received a single intravenous infusion of tedizolid phosphate dosed at 6 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
  Interventions: Drug: Tedizolid Phosphate (IV)
- Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 years) (Experimental): Participants 2 to <6 years of age received a single intravenous infusion of tedizolid phosphate dosed at 3 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
  Interventions: Drug: Tedizolid Phosphate (IV)
- Group 3: Tedizolid oral 4 mg/kg (6 to <12 years) (Experimental): Participants 6 to <12 years of age received a single dose of tedizolid phosphate oral suspension dosed at 4 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
  Interventions: Drug: Tedizolid Phosphate (oral suspension)
- Group 4: Tedizolid oral 3 mg/kg (2 to <6 years) (Experimental): Participants 2 to <6 years of age received a single dose of tedizolid phosphate oral suspension dosed at 3 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
  Interventions: Drug: Tedizolid Phosphate (oral suspension)

INTERVENTIONS:
Drug: Tedizolid Phosphate (IV) — 200 mg/vial powder for injection
  Other Names: Sivextro; TR-701 FA; MK-1986
  Arms: Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 years); Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 years); Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 years); Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 years)
Drug: Tedizolid Phosphate (oral suspension) — Powder for oral suspension 20 mg/mL following reconstitution
  Other Names: Sivextro; TR-701 FA; MK-1986
  Arms: Group 3: Tedizolid oral 4 mg/kg (6 to <12 years); Group 4: Tedizolid oral 3 mg/kg (2 to <6 years)

SUMMARY:
This is a study to assess the pharmacokinetics (PK) of tedizolid phosphate and its active metabolite, tedizolid, and the safety of tedizolid phosphate following administration of a single IV (Part A) or oral suspension (Part B) administration to hospitalized participants ages 6 to <12 years (Groups 1 and 3, respectively), and 2 to <6 years (Groups 2 and 4, respectively).

DETAILED DESCRIPTION:
Part A (IV):

* Group 1 (Cohort 1 and Cohort 2) (6 to <12 years)
* Group 2 (Cohort 1 and Cohort 2) (2 to <6 years)

Part B (Oral Suspension):

* Group 3 (6 to <12 years)
* Group 4 (2 to <6 years)

In Cohort 1 of Group 1 (IV) participants received a single administration of tedizolid phosphate at 5 mg/kg of total body weight. After all participants in Cohort 1 of Group 1 received study drug, a preliminary analysis of the safety and PK data was performed and results were used to select 4 mg/kg as the appropriate dose for Cohort 2 of Group 1 and Group 3, and to select 6 mg/kg as the starting dose for the younger participants, Cohort 1 of Group 2. After all participants in Cohort 1 of Group 2 receive study drug, another preliminary analysis of the safety and PK data will be performed and results will be used to confirm 6 mg/kg as the appropriate dose for Cohort 2 of Group 2. Similarly, the Group 4 dose will be confirmed after data review of Group 3 results.

ELIGIBILITY:
Inclusion Criteria:

* Receiving prophylaxis for or with a confirmed or suspected infection with Gram-positive bacteria and receiving concurrent antibiotic treatment with Gram-positive antibacterial activity;
* Weight >5th percentile and <95th percentile based on age;
* Stable condition as determined from medical history, physical examination, minimally 5-lead electrocardiogram (ECG), vital signs, and clinical laboratory evaluations;
* Females must be premenarchal, abstinent, or practicing an effective method of birth control;

Exclusion Criteria:

* History of seizures, other than febrile seizures, clinically significant cardiac arrhythmia, cystic fibrosis, moderate or severe renal impairment, or any physical condition that could interfere with the study results;
* Recent (3 month) history or current infection with viral hepatitis or other significant hepatic disease;
* History of drug allergy or hypersensitivity to oxazolidinones;
* Pregnant or breast feeding;
* Significant blood loss within 60 days prior to study start;
* Any acute or chronic condition that would limit the participant's ability to complete and/or participate in this clinical study.
* Treatment with investigational medicinal product within 30 days before the infusion/dose of study drug.
* Oral administration of methotrexate, topotecan, irinotecan or rosuvastatin, during administration of oral study drug. Administration during the follow-up period is allowed, as is administration during treatment with IV study drug.
* Use of monoamine oxidase inhibitors or serotonergic agents including tricyclic antidepressants, selective serotonin reuptake inhibitors, and serotonin 5 hydroxytryptamine receptor agonists (triptans), meperidine, or buspirone within,14 days prior to study, or planned use while on study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Arrieta AC, Ang JY, Espinosa C, Fofanov O, Tondel C, Chou MZ, De Anda CS, Kim JY, Li D, Sabato P, Sears PS, Bradley JS. Pharmacokinetics and Safety of Single-dose Tedizolid Phosphate in Children 2 to <12 Years of Age. Pediatr Infect Dis J. 2021 Apr 1;40(4):317-323. doi: 10.1097/INF.0000000000003030. PMID 33710976

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to enrollment, participants were receiving prophylaxis for or with a confirmed or suspected infection with gram-positive bacteria and receiving concurrent antibiotic treatment with gram-positive antibacterial activity.
Period: Overall Study
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Started | 5 | 5 | 5 | 5 | 6 | 6
Completed | 5 | 5 | 4 | 5 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.3) | 7.4 (1.1) | 3.4 (0.5) | 4.0 (1.4) | 8.5 (1.8) | 3.2 (1.0) | 5.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 2 | 4 | 13
  Male | 4 | 3 | 4 | 2 | 4 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 0 | 3 | 2 | 11
  Not Hispanic or Latino | 2 | 4 | 3 | 5 | 3 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 1 | 0 | 4
  White | 4 | 3 | 5 | 5 | 4 | 5 | 26
  More than one race | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Drug Concentration in Plasma (Cmax) of Tedizolid Phosphate (Prodrug)
Description: Cmax of tedizolid phosphate in participants ages 6 to <12 years (Group 1) and 2 to <6 years (Group 2). Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: IV: immediately after the end of the infusion, and various time points up to 48 hours after the start of infusion as described above. Oral: at various time points up to 48 hours after the dose as described above.
Population: All participants who received a dose of tedizolid phosphate and had at least one quantifiable (above the lower limit of quantification) post-administration concentration of tedizolid phosphate.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 4 | 5 | 5 | 4 | 6 | 1
ng/mL | 76.3 [8.38 to 695] | 82.4 [11.4 to 595] | 710 [98.4 to 5130] | 234 [25.7 to 2140] | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to report for this group. | 9.4 [NA to NA] — 95% CI cannot be calculated for a population containing only a single participant.

2. Primary Outcome: Time to Reach Peak Plasma Concentration (Tmax) of Tedizolid Phosphate (Prodrug)
Description: Time to reach peak plasma concentration (Tmax) of tedizolid phosphate in participants ages 6 to <12 years (Group 1) and 2 to <6 years (Group 2). Tedizolid phosphate concentrations were below the lower limit of quantification in Group 3 and Group 4. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 4 | 5 | 5 | 4 | 6 | 1
Hours | 1.18 [1.07 to 2.07] | 1.10 [1.00 to 1.33] | 1.12 [1.07 to 1.17] | 1.02 [1.00 to 1.05] | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to report for this group. | 6.0 [6.0 to 6.0]

3. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Tedizolid Phosphate (Prodrug) From Time Zero to Last Detectable Measurement
Description: Area under the plasma concentration time curve (AUC) of tedizolid phosphate from time zero to last detectable measurement following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid phosphate necessary to calculate the AUC.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 4 | 5 | 5 | 4 | 6 | 1
hr*ng/mL | 64.8 [6.42 to 654] | 63.6 [8.04 to 503] | 433 [54.8 to 3430] | 182 [18.1 to 1840] | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | 14.1 [NA to NA] — 95% CI cannot be calculated for a population containing only a single participant.

4. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Tedizolid Phosphate (Prodrug) From Time Zero to Infinity
Description: Area under the plasma concentration time curve (AUC) of tedizolid phosphate from time zero to infinity following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid phosphate necessary to calculate the AUC. Only 1 participant, from Group 2 Cohort 2, had analyzable data for this outcome measure.
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 1 | 6 | 6
hr*ng/mL | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | 2000 [2000 to 2000] | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA [NA to NA] — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group.

5. Primary Outcome: Terminal Elimination Half-life (T1/2) of Tedizolid Phosphate (Prodrug)
Description: Terminal elimination half-life (T1/2) of tedizolid phosphate following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid phosphate necessary to calculate the T1/2. Only 1 participant, from Group 2 Cohort 2, had analyzable data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 1 | 6 | 6
Hours | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | 2.77 (NA) — Geometric coefficient of variation cannot be calculated for a population containing only a single participant. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group.

6. Primary Outcome: Clearance (CL) of Tedizolid Phosphate (Prodrug) in Participants Who Received Tedizolid Phosphate Intravenously (IV)
Description: CL of IV tedizolid phosphate in participants ages 6 to <12 years (Group 1) and 2 to <6 years (Group 2).
Time Frame: Group 1 (6 to <12 years): Day 1 immediately after infusion and at 1.5, 2, 3, 4, 6, 12, and 24 hours. Group 2 (2 to <6 years): Day 1 immediately after infusion and at 3, 6, 12, 24 and 48 hours.
Population: All participants who received an IV infusion of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid phosphate necessary to calculate the CL. Only 1 participant, from Group 2 Cohort 2, had analyzable data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 1
mL/hr | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | 24400 (NA) — Geometric coefficient of variation cannot be calculated for a population containing only a single participant.

7. Primary Outcome: Clearance (CL/F) of Tedizolid Phosphate in Participants Who Received Oral Tedizolid Phosphate (Prodrug)
Description: CL/F of oral suspension tedizolid phosphate and its active metabolite, tedizolid, in participants ages 6 to <12 years (Group 3) and 2 to <6 years (Groups 4).
Time Frame: Group 3 (6 to <12 years): at 1, 2, 3, 4, 6, 8, 12, and 24 hours after the dose; Group 4 (2 to <6 years): at 3, 6, 9, 12, 24 and 48 hours after the dose
Population: All participants who received an oral dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid phosphate necessary to calculate the CL/F. All orally dosed participants' data were below the lower limit of quantification, resulting in no reportable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 6 | 6
mL/hr/kg | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group. | NA (NA) — All participants' results in this group were below the lower limit of quantification, so no data exist to present for this group.

8. Primary Outcome: Maximum Observed Drug Concentration in Plasma (Cmax) of Tedizolid (the Active Metabolite)
Description: Maximum observed drug concentration in plasma (Cmax) of tedizolid (active metabolite) following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had at least one quantifiable (above the lower limit of quantification) post-administration concentration of tedizolid.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 6
ng/mL | 4960 (3440) [3440 to 7140] | 4140 (2880) [2880 to 5970] | 7460 (5180) [5180 to 10800] | 4190 (2910) [2910 to 6030] | 2590 (1860) [1860 to 3620] | 1820 (1310) [1310 to 2550]

9. Primary Outcome: Time to Reach Peak Plasma Concentration (Tmax) of Tedizolid (the Active Metabolite)
Description: Time to reach peak plasma concentration (Tmax) of tedizolid (active metabolite) following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 6
Hours | 1.18 (1.07) [1.07 to 1.50] | 1.10 (1.00) [1.00 to 1.33] | 1.12 (1.07) [1.07 to 1.17] | 1.00 (1.00) [1.00 to 1.05] | 2.53 (1.20) [1.20 to 6.02] | 3.08 (3.00) [3.00 to 12.00]

10. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Tedizolid (Active Metabolite) From Time Zero to Last Detectable Measurement
Description: Area under the plasma concentration time curve (AUC) of tedizolid (active metabolite) from time zero to last detectable measurement following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid necessary to calculate the AUC.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 6
hr*ng/mL | 28200 (21200) [21200 to 37600] | 19700 (14800) [14800 to 26200] | 26800 (20200) [20200 to 35800] | 17100 (12800) [12800 to 22700] | 22700 (17500) [17500 to 29500] | 14600 (11200) [11200 to 18900]

11. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Tedizolid (Active Metabolite) From Time Zero to Infinity
Description: Area under the plasma concentration time curve (AUC) of tedizolid (active metabolite) from time zero to infinity following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5
hr*ng/mL | 29600 [22500 to 38900] | 21000 [16000 to 27600] | 27300 [20800 to 35900] | 17300 [13200 to 22700] | 24900 [19400 to 32000] | 17200 [13100 to 22600]

12. Primary Outcome: Terminal Elimination Half-life (T1/2) of Tedizolid (Active Metabolite)
Description: Terminal elimination half-life (T1/2) of tedizolid (active metabolite) following administration of IV or oral dose. Pharmacokinetic sampling occurred at the following time points: Group 1 (6 to <12 years): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (IV): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (6 to <12 years): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (2 to <6 years): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid necessary to calculate the T1/2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5
Hours | 5.18 (21.54) [lower limit 21.54] | 4.93 (13.82) [lower limit 13.82] | 5.51 (30.16) [lower limit 30.16] | 5.76 (29.20) [lower limit 29.20] | 6.15 (24.41) [lower limit 24.41] | 6.79 (10.85) [lower limit 10.85]

13. Primary Outcome: Clearance (CL) of Tedizolid (Active Metabolite) in Participants Who Received Tedizolid Phosphate Intravenously (IV)
Description: CL of IV tedizolid phosphate and its active metabolite, tedizolid, in participants ages 6 to <12 years (Group 1) and 2 to <6 years (Group 2).
Time Frame: as for outcome 6
Population: All participants who received an IV infusion of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid of tedizolid necessary to calculate the CL.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5
mL/hr | 4164.60 (36.39) | 4145.73 (73.21) | 2582.66 (20.64) | 2461.08 (11.99)

14. Primary Outcome: Clearance (CL/F) of Tedizolid (Active Metabolite) in Participants Who Received Oral Tedizolid Phosphate
Description: CL/F of tedizolid, in participants ages 6 to <12 years (Group 3) and 2 to <6 years (Groups 4).
Time Frame: as for outcome 7
Population: All participants who received an oral dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid of tedizolid necessary to calculate the CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 6 | 5
mL/hr/kg | 4073.32 (21.14) | 2090.77 (50.27)

15. Primary Outcome: Dose Normalized Area Under the Plasma Concentration Time Curve (AUC) of Tedizolid (Active Metabolite) From Time Zero to Infinity
Description: The area under the plasma concentration time curve (AUC) of tedizolid (active metabolite) from time zero to infinity following administration of IV or oral dose, normalized to dosage, was calculated. Per protocol, this outcome used pooled groups as follows: The IV Group pooled Groups 1 and 2, who received tedizolid phosphate via intravenous (IV) administration; the Oral Group pooled groups 3 and 4, who received tedizolid phosphate via oral administration. Pharmacokinetic sampling occurred at the following time points: Group 1 (part of the IV Group): Day 1 immediately after infusion and 1.5, 2, 3, 4, 6, 12, and 24 hours; Group 2 (part of the IV Group): Day 1 immediately after infusion and 3, 6, 12, 24 and 48 hours; Group 3 (part of the Oral Group): Day 1 at 1, 2, 3, 4, 6, 8, 12, and 24 hours after oral dose; Group 4 (part of the Oral Group): Day 1 at 3, 6, 9, 12, 24 and 48 hours after oral dose.
Time Frame: as for outcome 1
Population: All participants who received a dose of tedizolid phosphate and had adequate quantifiable (above the lower limit of quantification) post-administration concentrations of tedizolid necessary to calculate the AUC. Per protocol, participant arms were pooled based on route of administration (IV or Oral) and outcome was normalized to the dose received.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr*ng/mL/mg/kg
Groups:
- IV Group: Combined group of participants from Groups 1-2. Participants 2 to <12 years of age received a single intravenous infusion of tedizolid phosphate dosed at 3, 4, 5, or 6 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
- Oral Group: Combined group of participants from Groups 3-4. Participants 2 to <12 years of age received a single dose of tedizolid phosphate oral suspension dosed at 3 or 4 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
Arm/Group | IV Group | Oral Group
Number analyzed (Participants) | 20 | 11
hr*ng/mL/mg/kg | 5340 [4680 to 6100] | 6000 [5020 to 7180]
Statistical Analysis 1: Comparison: IV Group vs Oral Group; Test type: Other — Bioavailability: Geometric least squares mean ratio between the Oral Group's and IV Group's dose normalized AUC from time zero to infinity; Geometric Least Squares Mean Ratio = 1.12, 90% CI 2-sided [0.93 to 1.35] — The Oral Group represented the numerator in the bioavailability ratio, and the IV Group represented the denominator

16. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 9 days
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 6
Participants | 2 | 1 | 2 | 0 | 3 | 1

17. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 16
Time Frame: 1 day
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Palatability of Oral Tedizolid Phosphate Suspension in Participants Who Received Oral Tedizolid Phosphate
Description: Palatability of oral tedizolid phosphate suspension in participants ages 6 to <12 years (Group 3) and 2 to <6 years (Group 4). Palatability was assessed using a 5-point hedonic scale and spontaneous verbal judgment. This hedonic scale consists of 5 pictures of line drawn faces corresponding to very bad, bad, neither good nor bad, good and very good. The participant was asked to mark or point to the face to show how they felt about the taste of the study drug. For preverbal children, the score was assessed by the parent/caregiver, or study staff administering or witnessing administration of the study drug.
Time Frame: Following single oral dose on Day 1
Population: All participants who received an oral dose of tedizolid phosphate suspension.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (2 to <6 Years)
Number analyzed (Participants) | 6 | 6
Participants
  Very good | 0 | 0
  Good | 0 | 1
  Neither good nor bad | 3 | 2
  Bad | 1 | 3
  Very bad | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 9 days
Groups:
- Group 4: Tedizolid Oral 3 mg/kg (6 to <12 Years): Participants 2 to <6 years of age received a single dose of tedizolid phosphate oral suspension dosed at 3 mg/kg of total body weight. Maximum dose is 200 mg of tedizolid phosphate.
Arm/Group | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) | Group 4: Tedizolid Oral 3 mg/kg (6 to <12 Years)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5 | 2/5 | 0/5 | 3/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) (N=5) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) (N=5) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) (N=5) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) (N=5) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) (N=6) | Group 4: Tedizolid Oral 3 mg/kg (6 to <12 Years) (N=6)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Cohort 1: Tedizolid IV 5 mg/kg (6 to <12 Years) (N=5) | Group 1 Cohort 2: Tedizolid IV 4 mg/kg (6 to <12 Years) (N=5) | Group 2 Cohort 1: Tedizolid IV 6 mg/kg (2 to <6 Years) (N=5) | Group 2 Cohort 2: Tedizolid IV 3 mg/kg (2 to <6 Years) (N=5) | Group 3: Tedizolid Oral 4 mg/kg (6 to <12 Years) (N=6) | Group 4: Tedizolid Oral 3 mg/kg (6 to <12 Years) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to pursue publication of the results of the study in cooperation with a lead Investigator. Sponsor written approval is required for publication of any data subsets. Final authorship will be determined in accordance with the International Committee of Medical Journal Editors definition of authorship. Participant names and other personal data may not be disclosed in any publication without prior written authorization from Sponsor and the participant.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT02750761/Prot_SAP_000.pdf